CLINICAL TRIAL: NCT04299776
Title: A Randomized Clinical Trial on the Effects of Active Intrathoracic Pressure Regulation Therapy on Hemodynamic Stability During Shoulder Surgery in the Sitting Position
Brief Title: CirQPOD Shoulder Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Review of new pre-clinical data
Sponsor: Zoll Medical Corporation (Industry)
Collaborators: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 40701
Record Dates: First submitted 2020-03-02; First posted 2020-03-09 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Hypotension on Induction
Keywords: Intraoperative hypotension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- IPR therapy (Experimental): Intrathoracic pressure regulation (IPR) therapy level of -10 cmH2O (-7 cmH2O for run-in) provided by the CirQPOD device during shoulder surgery in the sitting position
  Interventions: Device: CirQPOD
- Standard airway (Active Comparator): Standard airway pressure (PEEP of +5 cmH2O) during shoulder surgery in the sitting position
  Interventions: Device: Standard airway management

INTERVENTIONS:
Device: CirQPOD — CirQPOD is connected between the wye piece on ventilator/anesthesia machine tubing and the patient's airway and generates negative intrathoracic pressure during the expiratory phase of ventilation which has been shown to improve blood flow.
  Arms: IPR therapy
Device: Standard airway management — Standard airway management during surgery (PEEP of +5 cmH2O)
  Arms: Standard airway

SUMMARY:
Intrathoracic pressure regulation (IPR) therapy, delivered by impedance threshold devices (ITDs) or intrathoracic pressure regulators (ITPRs), increases venous return, preload, cardiac output, blood pressure, and cerebral perfusion pressure by intermittently creating negative intrathoracic pressure, which improves circulation in hypotensive animals and humans. By increasing systemic pressure and cerebral perfusion as well as promoting venous return, IPR therapy potentially improves cerebral oxygenation. The lower intrathoracic pressures may also reduce pulmonary artery pressure, although there is currently little evidence one way or the other. Use of an ITPR can counteract the multifactorial intraoperative hypotension common during surgeries under general anesthesia, and reduce the need for other measures to treat such hypotension; however, they might simultaneously promote pulmonary complications.

The investigators will therefore assess whether the use of intrathoracic pressure regulation in adults having shoulder surgery under general anesthesia in the sitting position reduces vasoactive medication requirements compared with routine clinical practice. Simultaneously, the investigators will assess the effect of intrathoracic pressure regulation on pulmonary circulation, cerebral oxygenation, and postoperative atelectasis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* American Society of Anesthesiologists (ASA) physical status class ≤3
* Scheduled for surgery in sitting/ beach-chair positions under general anesthesia in the Cleveland Clinic main campus
* Planned length of surgery >60 minutes

Exclusion Criteria:

* Severe peripheral vascular disease or other contraindication for use of vasopressor infusion
* Obstructive lung disease - moderate or severe asthma or COPD
* Baseline hypoxemia (SpO2<92% on room air)
* Body Mass Index (BMI) >35
* Congestive heart failure
* Pneumothorax or hemothorax
* Uncontrolled hemorrhage
* Planned intraoperative hypotension
* Contraindication to trans-esophageal echocardiography (esophageal stricture, surgery involving the esophagus or stomach)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01-28 (Actual); Primary Completion 2020-03-28 (Actual); Study Completion 2020-03-28 (Actual)

PRIMARY OUTCOMES:
Phenylephrine use | from device placement to start of wound closure, a period of up to four hours
  Amount of phenylephrine required to maintain MAP of 80±5 mmHg

SECONDARY OUTCOMES:
Pulmonary artery pressure | at least two minutes after IPR level of -10 cmH2O has been set
  pressure in the pulmonary artery as measured by transesophageal echocardiography (TEE)
Atelectasis | first day post-op
  presence and amount of atelectasis as determined by chest computerized tomography (CT)
PaO2 | at least 20 minutes, but not more than 2 hours, after patient is free of oxygen supplementation
  post-operative partial arterial oxygen pressure measured by arterial blood gas (ABG)

CONTACTS AND LOCATIONS:
Locations (1):
- Outcomes Research, Anesthesia Institute, Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No